CLINICAL TRIAL: NCT00328718
Title: Randomised, Double-blind, Double-dummy, Parallel-group, Comparative Study of Salmeterol/FP 50/100mcg bd Inhalation Powder Via Diskus With Oral Montelukast (5mg QD) Chewable Tablets in Children 6-14 Years
Brief Title: Pediatric ADVAIR DISKUS Versus Oral Montelukast Chewable Tablets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM103848
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Asthma
Keywords: Persistent Asthma; pediatric asthmatic; asthma control
MeSH Terms: conditions — Asthma | interventions — montelukast; Salmeterol Xinafoate; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: montelukast (5mg QD)
Drug: Salmeterol/Fluticasone propionate Inhalation Powder (50/100mcg BID)
  Other Names: montelukast (5mg QD)

SUMMARY:
This study is being conducted to demonstrate the superior clinical effectiveness of Salmeterol/Fluticasone Propionate compared to montelukast in the management of persistent asthma in children aged 6-14 years, and to assess the effect of each treatment [Salmeterol/Fluticasone Propionate (50/100 mcg) and montelukast (5 mg)] on lung function, asthma control, Health Outcomes including the child's quality of life as measured by Paediatric Asthma Quality of Life Questionnaire (PAQLQ) and the caregiver's quality of life as measured by Paediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) at selected centers where a valid translation is available.

DETAILED DESCRIPTION:
Pediatric Asthma Clinical Effectiveness study (PEACE). A Randomized, Double-Blind, Double Dummy, Parallel Group comparative clinical study of Salmeterol/Fluticasone propionate Inhalation Powder (50/100mcg BID) via DISKUS† with Oral montelukast (5mg QD) Chewable Tablets in Children 6-14 years of Age with Persistent Asthma

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of asthma for at least 6 months (per American Thoracic Society [ATS] definition).
* Best forced expiratory volume in one second (FEV1) between 55% and 80% of predicted normal.
* More than or 12% FEV1 reversibility following inhalation of salbutamol.
* Must also be symptomatic on short-acting beta-agonists.
* Must not have used inhaled corticosteroids over the previous month or LTRAs (Leukotriene antagonists)over the previous 2 weeks.

Exclusion criteria:

* Hospital admission for asthma within 3 months prior to Visit 1.
* Sinus, middle ear, oropharyngeal, upper or lower respiratory tract infections within two weeks immediately preceding Screening Visit 1.
* Oral or parenteral steroid therapy in the last 12 weeks, or more than 3 courses in the last 6 months.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 526
Dates: Start 2005-10 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean morning PEFR (Peak Expiratory Flow Rate) at endpoint.

SECONDARY OUTCOMES:
Changes from baseline to endpoint of:morning pre-dose FEV1 (Forced expiratory volume) symptom free 24 hour-periods rescue medication-free 24 hour-periods mean evening PEFR

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- Argentina (3):
  - GSK Investigational Site, Santa Fe, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal-Buenos Aires
- Colombia (3):
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Cali
  - GSK Investigational Site, Medellín
- GSK Investigational Site, San José, Costa Rica
- Mexico (5):
  - GSK Investigational Site, Chihuahua City, Chihuahua
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- GSK Investigational Site, Lima, Lima Province, Peru
- Turkey (Türkiye) (6):
  - GSK Investigational Site, Adana
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Antalya
  - GSK Investigational Site, Bursa
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir
- GSK Investigational Site, Caracas, Venezuela

REFERENCES:
- [Background] Maspero J, Guerra F, Cuevas F, Gutierrez JP, Soto-Ramos M, Anderton S, Mechali D, Chan R, Pedersen S. Efficacy and tolerability of salmeterol/fluticasone propionate versus montelukast in childhood asthma: A prospective, randomized, double-blind, double-dummy, parallel-group study. Clin Ther. 2008 Aug;30(8):1492-504. doi: 10.1016/j.clinthera.2008.07.018. PMID 18803991